CLINICAL TRIAL: NCT02423057
Title: Phase I Trial of 4'-Thio-2'-Deoxycytidine (TdCyd) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150116; 15-C-0116
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Neoplasms; Solid Tumors
Keywords: Pharmacodynamics; DNA Methylation; Pharmacokinetics; Nucleoside Analog; Epigenetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): TdCyd will be administered orally once a day for 5 days of each week for 2 weeks, with one week off, in 21-day cycles
  Interventions: Drug: TdCyd

INTERVENTIONS:
Drug: TdCyd — Methylation-mediated silencing of genes is an epigenetic mechanism implicated in carcinogenesis; agents that inhibit this mechanism are of clinical interest because of their potential to re-activate silenced tumor suppressor genes. The nucleoside analog 4'-thio-2'-deoxycytidine (TdCyd) is incorporated into DNA where it engages the active site of DNA methyltransferase I (DNMT1), a maintenance methyltransferase that contributes to the hypermethylation and silencing of tumor suppressor genes. TdCyd offers an improvement over current DNMT inhibitors by virtue of a higher incorporation rate into DNA at lower levels of cytotoxicity; treatment with TdCyd is anticipated to result in the inhibition of tumor growth due to DNMT1 depletion at oral doses that are well tolerated in extended dosing schedules.

SUMMARY:
Background:

- Genes are made up of DNA and are the instruction book for cells. When people have cancer, some of the genes that might have slowed the growth of tumor cells were turned off. Researchers think a drug called TdCyd might help to turn these genes back on. This may slow the growth of tumors in people with cancer.

Objectives:

- To test the safety of TdCyd and to find out how it works. Also, to find out the dose of the drug that can be safely given to humans.

Eligibility:

- Adults 18 years and older who have advanced cancer that has progressed after standard treatment, or for which no effective therapy exists.

Design:

* Participants will take TdCyd by mouth. The drug is given in 21-day cycles. TdCyd is taken once a day during week 1 for 5 days. Then for 2 days participants do not take the drug. Then they take it for 5 days during week 2. No TdCyd is taken during week 3.
* Participants will keep a diary of their study drug doses.
* Participants will have tests about every 3 weeks to see how the study drugs are affecting their body. They will have blood and urine tests, a medical history, and physical exams. They may have computed tomography (CT) scans to measure their tumors. They may have an electrocardiogram, which measures the heart electrical activity.
* If participants develop any side effects, they may be asked to visit more often.
* Participants will stay in the study as long as they are tolerating TdCyd and their tumors are either stable or getting better. One month after stopping the drug, they will have a follow-up phone call.

DETAILED DESCRIPTION:
Background:

* Methylation-mediated silencing of genes is an epigenetic mechanism implicated in carcinogenesis; agents that inhibit this mechanism are of clinical interest because of their potential to re-activate silenced tumor suppressor genes. Two DNA hypomethylating nucleosides, 5-azacytidine (azacytidine) and 5-aza-2'-deoxycytidine (decitabine) have been approved by the FDA for the treatment of patients with myelodysplastic syndromes and certain leukemias.
* The nucleoside analog 4'-thio-2'-deoxycytidine (TdCyd) is incorporated into DNA where it engages the active site of DNA methyltransferase I (DNMT1), a maintenance methyltransferase that contributes to the hypermethylation and silencing of tumor suppressor genes. DNMT1 can become trapped in a covalent complex with DNA, thus depleting free enzyme and inhibiting the normal maintenance methylation of CpG sites, resulting in reactivation of tumor suppressor genes.
* Data generated at Southern Research Institute and the NCI suggest a correlation between TdCyd activity in solid tumor xenograft models and decreased levels of DNMT1.
* TdCyd offers an improvement over current DNA methyltransferase inhibitors by virtue of a higher incorporation rate into DNA at lower levels of cytotoxicity; treatment with TdCyd is anticipated to result in the inhibition of tumor growth due to DNMT1 depletion at oral doses that are well tolerated in extended dosing schedules.
* Two patients on dose levels 6 and 7 developed Pneumocystis jiroveci pneumonia (PJP) so all patients will be administered PJP prophylaxis.

Primary Objective:

-To establish the safety, tolerability, and MTD of oral TdCyd administered daily for 5 days a week for 2 weeks, with one week off, q 21-day cycles, to patients with refractory solid tumors

Secondary Objectives:

* To determine the pharmacokinetics of oral TdCyd
* To document preliminary evidence of TdCyd activity
* To determine effect of study treatment on re-expression of select genes silenced by methylation in circulating tumor cells

Eligibility:

-Patients must have histologically documented solid tumors whose disease has progressed on standard therapy or for which there is no available standard therapy

Study Design:

* TdCyd will be administered orally once a day for 5 days of each week for 2 weeks, with one week off, in 21-day cycles.
* The trial will follow an accelerated titration design, changing to a traditional 3+3 dose escalation design (3-6 patients per cohort) once specified toxicity criteria are met. Intrapatient dose escalation will be allowed.
* Blood samples will be obtained for pharmacokinetic analysis and to isolate circulating tumor cells to assess re-expression of genes silenced by methylation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented solid tumors whose disease has progressed on standard therapy or for which there is no available standard therapy.
* Patients must have measurable or evaluable disease.
* Age greater than or equal to 18 years of age.
* ECOG performance status less than or equal to 2.
* Life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

  1. absolute neutrophil count greater than or equal to 1,500/mcL
  2. platelets greater than or equal to 100,000/mcL
  3. total bilirubin less than or equal to 1.5 times institutional upper limit of normal
  4. AST(SGOT)/ALT(SGPT) less than or equal to 3 times institutional upper limit of normal
  5. creatinine less than or equal to 1.5 times institutional upper limit of normal

OR

e. creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above 1.5 times institutional normal

* Because nucleoside analogs are known to be teratogenic, women of child-bearing potential and men must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence; sterilization) prior to study entry, for the duration of study participation, and for 3 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use two forms of contraception prior to the study, for the duration of study participation, and for 3 months after completion of administration of TdCyd.
* Patients must have completed any chemotherapy, radiation therapy, or biologic therapy greater than or equal to 4 weeks or 5 half-lives (whichever is shorter) (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a phase 0 or equivalent study and be greater than or equal to 2 weeks since any prior palliative radiation or cyberknife therapy. Patients must have recovered to grade 1 from prior toxicity or adverse events. Patients with bone metastases or hypercalcemia on intravenous bisphosphonate treatment prior to study entry may continue this treatment.
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to provide blood and urine samples for research purposes.
* Ability to swallow pills/capsules.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Pregnant women and women who are breastfeeding are excluded from this study.
* Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to active or uncontrolled infection, immune deficiencies, known HIV infection requiring protease inhibitor therapy, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 1 month after treatment of the brain metastases. Patients should not be on anti-seizure medications. These patients may be enrolled at the discretion of the Principal Investigator.
* Malabsorption syndrome or other conditions that would interfere with intestinal absorption.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, and MTD of oral TdCyd administered daily for 5 days a week for 2 weeks, with one week off, q 21-day cycles | Cycle 1
  To determine the safety, tolerability, and MTD of oral TdCyd administered daily for 5 days a week for 2 weeks, with one week off, q 21-day cycles

SECONDARY OUTCOMES:
To document preliminary evidence of TdCyd activity | Cycle 1 and 2
  To document preliminary evidence of TdCyd activity (using RECIST criteria)

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cowan LA, Talwar S, Yang AS. Will DNA methylation inhibitors work in solid tumors? A review of the clinical experience with azacitidine and decitabine in solid tumors. Epigenomics. 2010 Feb;2(1):71-86. doi: 10.2217/epi.09.44. PMID 22122748
- [Background] Thottassery JV, Sambandam V, Allan PW, Maddry JA, Maxuitenko YY, Tiwari K, Hollingshead M, Parker WB. Novel DNA methyltransferase-1 (DNMT1) depleting anticancer nucleosides, 4'-thio-2'-deoxycytidine and 5-aza-4'-thio-2'-deoxycytidine. Cancer Chemother Pharmacol. 2014 Aug;74(2):291-302. doi: 10.1007/s00280-014-2503-z. Epub 2014 Jun 8. PMID 24908436
- [Background] Kumar S, Horton JR, Jones GD, Walker RT, Roberts RJ, Cheng X. DNA containing 4'-thio-2'-deoxycytidine inhibits methylation by HhaI methyltransferase. Nucleic Acids Res. 1997 Jul 15;25(14):2773-83. doi: 10.1093/nar/25.14.2773. PMID 9207024
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0116.html